CLINICAL TRIAL: NCT00562302
Title: A Prospective, Randomized, Multi-centered Safety and Efficacy Evaluation of the Bio-Seal Track Plug for Reducing Pneumothorax Rates Post Lung Biopsy
Brief Title: Bio-Seal Biopsy Track Plug for Reducing Pneumothorax Rates Post Lung Biopsy Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Angiotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BS-1053
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Pneumothorax
Keywords: lung biopsy
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-Seal Group (Experimental): Bio-Seal Plug Implanted
  Interventions: Device: Bio-Seal Plug
- Control Group (No Intervention): Control group with no intervention

INTERVENTIONS:
Device: Bio-Seal Plug — Deployment of the Bio-Seal plug in needle track
  Other Names: Bio-Seal™ Lung Biopsy Tract System
  Arms: Bio-Seal Group

SUMMARY:
BS-1053 A Prospective Randomized Multi-Centered Safety and Efficacy Evaluation of the Bio-Seal Biopsy Track Plug for Reducing Pneumothorax Rates Post Lung Biopsy Procedures

DETAILED DESCRIPTION:
This is a multi-centered, randomized trial in patients receiving lung biopsies. Patients will be randomized to either receive or not receive a Bio-Seal Biopsy Track Plug after a lung biopsy per standard hospital protocol. This study is designed to demonstrate safety and efficacy of the Bio-Seal Biopsy Track Plug in reducing pneumothorax rates post lung biopsy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must meet all medical conditions for lung biopsy;
* The patient must be at least 18 years of age;
* The patient, or legal representative, must understand and provide written consent for the procedure;
* The patient has a non-calcified, radiologically suspicious opacity or lung nodule, including a metastatic lung module, or mass of at least 1.0 cm in size; as determined by CT scan equipped with measurement software. Suspicious nodules observed by CT scan are defined as non-calcified masses with convex borders, not known to be stable. Suspicious nodules can also be defined as masses demonstrating opacity on chest x-ray that are suspicious by radiographic or clinical means and require biopsy.

Exclusion Criteria:

* Patients with radiological findings of bullous emphysema located in the area of the anticipated biopsy and biopsy needle track;
* Patients who cannot tolerate mild sedation, possibly secondary to poor respiratory status;
* Female patients who are pregnant. Note: patients of childbearing potential must have a serum or urine pregnancy test no more than one week prior to the biopsy procedure, and be instructed not to have unprotected sexual intercourse after the test until the biopsy procedure is completed.
* Patients who are uncooperative or cannot follow instructions.
* Patients who are currently enrolled in another IDE or IND clinical investigation that has not completed the required follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Director — Angiotech Pharmaceuticals
Locations (18):
- United States (18):
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - St. Josephs Radiology Limited, Tuscon, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Univerisity of California, San Diego, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Vascular and Interventional Radiology, New Haven, Connecticut
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Florida Research Network, Gainesville, Florida
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - St. Louis Medical Center, St Louis, Missouri
  - Univeristy of Cincinnati Medical Center, Cincinnati, Ohio
  - St Lukes Hospital, Bethlehem, Pennsylvania
  - Memorial Medical Center, Johnstown, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baptist Memorial Hospital, Memphis, Tennessee
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Evergreen Healthcare Diagnostic Imaging, Kirkland, Washington
  - Sacred Heart Medical Center & Heart Institute of Spokane, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bio-Seal Group | Control Group
Started | 170 | 169
Completed | 150 | 137
Not Completed | 20 | 32
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 0 | 6
Not completed — Non-compliance | 1 | 2
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Death | 1 | 2
Not completed — Lung resection prior to study completion | 7 | 7
Not completed — Not stated | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bio-Seal Group | Control Group | Total
Number analyzed (Participants) | 170 | 169 | 339
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (11.47) | 67.2 (12.38) | 66.7 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 75 | 167
  Male | 78 | 94 | 172
History of Smoking [Number; unit: Participants]
  Yes | 145 | 146 | 291
  No | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Treatment Success
Description: Treatment success was defined as the absence of a pneumothorax at each of the three follow-up time periods (0-60 minutes, 24 hours and 30 days).
Time Frame: 30 days
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 150 | 137
participants | 126 | 94

2. Secondary Outcome: Incidence of Chest Tube Placement
Description: A chest tube is the definitive initial treatment of a pneumothorax.
Time Frame: 30 days
Population: Intent to treat Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 6 | 18

3. Secondary Outcome: Time to Ambulation
Time Frame: 30 days
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
Hours | 3.3 (4.63) | 3.8 (6.29)

4. Secondary Outcome: Incidence of Hospital Admissions for Pneumothorax
Time Frame: 30 day
Population: Intent to treat Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 16 | 23

5. Secondary Outcome: Incidence of Adverse Events Related to the Procedure and Device Effects
Description: Anticipated, device-related adverse events that were defined in the original protocol.
Time Frame: 30 Day
Population: Intent to Treat Patients
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 43 | 74

6. Secondary Outcome: Number of Participants With Additional Chest X-rays Needed
Time Frame: 30 day
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 29 | 52

7. Secondary Outcome: Participants Discharged Beyond Hospital's Standard of Care
Description: Current standard of care for hospital discharge varies. Some institutions allow the patient to be discharged after a 3 hour wait. Others allow discharge after an x-ray indicates no pneumothorax. Since this study was randomized with control patients, the time to discharge beyond the hospital's standard of care was recorded to see if a trend for later discharge was apparent. This measure indicates the number of participants who were discharged later than their hospital's standard of care.
Time Frame: 30-day
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 8 | 18

8. Secondary Outcome: Incidence of Adverse Events
Description: Any treatment emergent adverse events (not considered device related by the investigators).
Time Frame: 30 days
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Bio-Seal Group | Control Group
Number analyzed (Participants) | 170 | 169
participants | 31 | 36

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Bio-Seal Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/170 | 2/169
Other Adverse Events (participants affected / at risk) | 60/170 | 90/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bio-Seal Group (N=170) | Control Group (N=169)
PULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SYNCOPE (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bio-Seal Group (N=170) | Control Group (N=169)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 9 (9)
VOMITING (Gastrointestinal disorders) | 5 (5) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
STOMATITIS (General disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 2 (2)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CHEST PAIN (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
PYREXIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
ENERGY INCREASED (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
INFUSION SITE PAIN (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PUNCTURE SITE PAIN (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAEMOTHORAX (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 0 (0) | 1 (1)
Allergic reaction to anesthesia/drugs (Immune system disorders) | 0 (0) | 1 (1) — Anticipated Adverse Device Effect
Bleeding at puncture site (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Anticipated Adverse Device Effect
Emphysema (subcutaneous) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Anticipated Adverse Device Effect
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) — Anticipated Adverse Device Effect
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 53 (53) — Anticipated Adverse Device Effect
Pleural fluid (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) — Anticipated Adverse Device Effect
Chest pain with pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (13) — Anticipated Adverse Device Effect
Chest pain without pneumothorax (Cardiac disorders) | 9 (11) | 11 (11) — Anticipated Adverse Device Effect
Puncture site bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Anticipated Adverse Device Effect
Fatigue (General disorders) | 0 (0) | 1 (1) — Anticipated Adverse Device Effect
Coughing with Blood (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) — Anticipated Adverse Device Effect
Altered lung function (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Anticipated Adverse Device Effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No